CLINICAL TRIAL: NCT01550068
Title: A Population-Based Study of Prevalence of Rheumatic Heart Disease and Cardiovascular Outcomes Among Schoolchildren in Nepal
Brief Title: Rheumatic Heart Disease School Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Thomas Pilgrim, MD, Department of Cardiology, Bern University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 018/12
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Rheumatic Heart Disease
Keywords: Rheumatic Heart Disease
MeSH Terms: conditions — Rheumatic Heart Disease | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Arm (Experimental): Echocardiographic screening
  Interventions: Diagnostic Test: Echocardiography
- Control Arm (No Intervention): No echocardiographic screening

INTERVENTIONS:
Diagnostic Test: Echocardiography
  Arms: Experimental Arm

SUMMARY:
Acute rheumatic Fever (ARF) results from an autoimmune response due to molecular mimicry between the M-protein on the group A β-hemolytic streptococci (GABHS) cell membrane and cardiac myosin, and may lead through recurrent or sustained inflammation to Rheumatic Heart Disease (RHD). RHD remains a major contributor to morbidity and premature death in the working age population in Nepal. Secondary prevention with regular oral or intravenous administration of penicillin continued until early adulthood is recommended to prevent the progression of the development of endocarditis and subsequent valvular dysfunction.

Screening for rheumatic heart disease using echocardiography has the potential to detect rheumatic valvular lesions at an earlier, clinically silent stage, as compared to clinical examination alone and might have a beneficial impact on long-term outcome of children with RHD. Schoolchildren aged 5-16 years from several public and private schools from rural and urban areas in Southeastern Nepal will be screened for RHD using portable echocardiography.

Three main inter-related objectives will be pursued in three phases of the study: In a first phase using a cross sectional approach, the prevalence of clinical and subclinical RHD will be investigated among a representative sample of schoolchildren from public and private schools in urban and rural areas. In a second phase, using a cohort study approach among those children diagnosed at different stages of RHD, clinical outcomes with regular medical surveillance will be assessed (a), and clinical and social risk factors associated with prognosis of the disease after receiving medical care at various stages of disease at diagnosis will be determined (b). A third phase will integrate the prevalence rates from phase 1 and the clinical outcomes from phase 2 in a mathematical model to assess the impact of screening and RHD treatment on health resource utilization.

DETAILED DESCRIPTION:
Background

Acute rheumatic Fever (ARF) results from an autoimmune response due to molecular mimicry between the M-protein on the group A β-hemolytic streptococci (GABHS) cell membrane and cardiac myosin, and may lead through recurrent or sustained inflammation to Rheumatic Heart Disease (RHD) (1). RHD is reported to affect over 15 million people worldwide and remains a major contributor to morbidity and premature death in the working age population in developing countries (2). Socioeconomic determinants such as poverty, overcrowding, and malnutrition have been related to RHD. The prevalence of ARF and RHD seems to be particularly high in Southeast Asia, the Western Pacific and Africa (3). Whereas heart murmurs detected on clinical examination may indicate clinically manifest RHD, echocardiographic screening revealed ten times higher prevalence rates of RHD among schoolchildren (4) and may help diagnose RHD at an earlier, "clinically silent" stage.

Patients with a past medical history of ARF or RHD are recommended secondary prevention with regular oral or intravenous administration of penicillin continued until early adulthood.

Even though preventive measures with penicillin are inexpensive and efficient, this strategy is difficult to effectuate in developing countries with limited access to health care resources.

A recent study proved that enrolling patients with ARF and RHD in a registry with close follow-up increases compliance to treatment and thus helps in reducing the cardiovascular sequelae associated with disease progression (5).

The prevalence of RHD among schoolchildren in urban and rural areas in Nepal is largely unknown, and risk factors associated with prognosis of the disease after receiving medical care at various stages of disease at diagnosis need to be determined. Moreover, the impact of screening using echocardiography, detecting RHD at an earlier, "clinically silent" stage of RHD on health resource utilization has to be determined.

Objective

Originally, three main inter-related objectives were to be pursued in three phases of the study: In the first phase using a cross sectional approach, the prevalence of clinical and subclinical RHD were to be investigated among a representative sample of schoolchildren from public and private schools in urban and rural areas. In the second phase, using a cohort study approach among those children diagnosed at different stages of RHD, clinical outcomes with regular medical surveillance were to be assessed (a), and clinical and social risk factors associated with prognosis of the disease after receiving medical care at various stages of disease at diagnosis were to be determined (b). A third phase was to integrate the prevalence rates from phase 1 and the clinical outcomes from phase 2 in a mathematical model to assess the impact of screening and RHD treatment on quality of life and health resource utilization.

On August 14 2013, the Nepal Health Research Council required the introduction of a control group in the design of the Rheumatic Heart Disease (RHD) School Project. The original design included a random sampling stratified by urban versus rural location and public versus private status of schools, with a computer-generated random sequence used to determine which schools would be centrally selected during Phase 1 of the project to undergo screening for RHD. The original computer-generated random sequence was therefore used to determine which schools would be randomly selected as control schools which did not undergo the screening intervention during Phase 1, but would be selected for follow-up during Phase 2 of the project. This approach implicitly allowed for a cluster randomized comparison between intervention and control schools at follow-up in children aged 5 to 12 years at baseline, when phase 1 of the study took place.

Methods

The project will employ three types of study designs performed in sequential phases: a cross sectional study (part 1), a longitudinal cohort study (part 2) and an analysis of the impact of screening, secondary prevention and treatment on health resource utilization (part 3).

1. Part 1: Cross-Sectional Survey Schoolchildren aged 5-16 years will be screened at selected schools in the Southeast area of Nepal. A follow-up examination will be performed in a subset of schools that underwent screening at baseline and in all control schools, allowing for a cluster randomized comparison at follow-up between schools that underwent screening at baseline and control schools in children aged 5 to 12 years at baseline.
2. Part 2: Longitudinal Cohort Study Those children with documented history of ARF and/or RHD will be included into a prospective registry and receive secondary prevention will be followed on a regular basis.
3. Part 3: Impact of Screening and Treatment of RHD The third phase will integrate the prevalence rates from phase 1 and the clinical outcomes from phase 2 in a mathematical model to assess the impact of screening and RHD treatment on health resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren in Southeast Nepal aged 5-16 years
* Written informed consent by the principal of the school
* Passive consent from the parents

Exclusion Criteria

* No formal exclusion criteria apply

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8519 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Rheumatic Heart Disease | 12 Months Screening Period

SECONDARY OUTCOMES:
composite of all-cause mortality, stroke, endocarditis, hospitalization for congestive heart failure, valvular surgery, mitral balloon valvuloplasty, and recurrence of rheumatic fever | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pilgrim, MD, Principal Investigator — Department of Cardiology, Bern University Hospital, Switzerland; Nikesh R Shrestha, MD, FESC, Principal Investigator — Department of Internal Medicine and Cardiology, B.P. Koirala Institute of Health Sciences (BPKIHS)
Locations (1):
- Department of Internal Medicine and Cardiology, B.P. Koirala Institute of Health Sciences (bpkihs), Dharan, Nepal

REFERENCES:
- [Background] Sadiq M, Islam K, Abid R, Latif F, Rehman AU, Waheed A, Azhar M, Khan JS. Prevalence of rheumatic heart disease in school children of urban Lahore. Heart. 2009 Mar;95(5):353-7. doi: 10.1136/hrt.2008.143982. Epub 2008 Oct 24. PMID 18952636
- [Background] Carapetis JR, McDonald M, Wilson NJ. Acute rheumatic fever. Lancet. 2005 Jul 9-15;366(9480):155-68. doi: 10.1016/S0140-6736(05)66874-2. PMID 16005340
- [Background] Seckeler MD, Hoke TR. The worldwide epidemiology of acute rheumatic fever and rheumatic heart disease. Clin Epidemiol. 2011 Feb 22;3:67-84. doi: 10.2147/CLEP.S12977. PMID 21386976
- [Background] Marijon E, Celermajer DS, Tafflet M, El-Haou S, Jani DN, Ferreira B, Mocumbi AO, Paquet C, Sidi D, Jouven X. Rheumatic heart disease screening by echocardiography: the inadequacy of World Health Organization criteria for optimizing the diagnosis of subclinical disease. Circulation. 2009 Aug 25;120(8):663-8. doi: 10.1161/CIRCULATIONAHA.109.849190. Epub 2009 Aug 10. PMID 19667239
- [Background] Pelajo CF, Lopez-Benitez JM, Torres JM, de Oliveira SK. Adherence to secondary prophylaxis and disease recurrence in 536 Brazilian children with rheumatic fever. Pediatr Rheumatol Online J. 2010 Jul 26;8:22. doi: 10.1186/1546-0096-8-22. PMID 20659324
- [Derived] Shrestha NR, Bruelisauer D, Uranw S, Mahato R, Sherpa K, Agrawal K, Rothenbuhler M, Karki P, Pilgrim T. Mid-term outcome of children with latent rheumatic heart disease in eastern Nepal. Open Heart. 2021 Apr;8(1):e001605. doi: 10.1136/openhrt-2021-001605. PMID 33820851
- [Derived] Karki P, Uranw S, Bastola S, Mahato R, Shrestha NR, Sherpa K, Dhungana S, Odutayo A, Gurung K, Pandey N, Agrawal K, Shah P, Rothenbuhler M, Juni P, Pilgrim T. Effectiveness of Systematic Echocardiographic Screening for Rheumatic Heart Disease in Nepalese Schoolchildren: A Cluster Randomized Clinical Trial. JAMA Cardiol. 2021 Apr 1;6(4):420-426. doi: 10.1001/jamacardio.2020.7050. PMID 33471029
- [Derived] Pilgrim T, Kalesan B, Karki P, Basnet A, Meier B, Urban P, Shrestha NR. Protocol for a population-based study of rheumatic heart disease prevalence and cardiovascular outcomes among schoolchildren in Nepal. BMJ Open. 2012 Jun 8;2(3):e001320. doi: 10.1136/bmjopen-2012-001320. Print 2012. PMID 22685225